CLINICAL TRIAL: NCT06353178
Title: BEACON Study: Virtual Coping Skills Groups for Cancer Patients, Survivors and Their Caregivers
Brief Title: Building Empowerment and Coping Outcomes for CaNcer Patients, Survivors and Their Caregivers
Acronym: BEACON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Color Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20240314
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Caregiving Stress; Caregiver Burnout; Survivorship
Keywords: cancer; caregiving; emotional support; psychology
MeSH Terms: conditions — Neoplasms; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to waitlist or intervention group. Those in intervention group will receive the peer program; those on the waitlist will receive it after being on the waitlist for 3 months.
Masking Description: Participants will be notified of a waitlist assignment upon enrolling. Those on the waitlist will receive the intervention after 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer Connect Program (Experimental): Participants assigned to this arm will be able to attend the online peer program upon entering the study.
  Interventions: Behavioral: Cancer Connect Program
- Waitlist (Placebo Comparator): Participants assigned to this arm will be on a waitlist and will be invited to join the online peer program in 3 months.
  Interventions: Behavioral: Cancer Connect Program

INTERVENTIONS:
Behavioral: Cancer Connect Program — Online group peer program where participants learn evidence based skills for managing stressors and emotions related to their cancer experience.

SUMMARY:
Cancer has a psychological, emotional and social impact beyond a patient's physical health. This study examines three new online peer mental-wellness support program for cancer patients, survivors or their caregivers. Each program teaches evidence-based skills, in the context of that groups lived experience, to manage the emotional impact of cancer. This study examines the impact of that program.

DETAILED DESCRIPTION:
Cancer has a psychological, emotional and social impact beyond a patient's physical health. These problems often ripple beyond the individual with the diagnosis, to their broader community, and also beyond a cancer treatment course into survivorship. As a result, there are a wide range of socioemotional needs in those who have been impacted by cancer. Further, these emotional impacts have a direct impact on morbidity and mortality of cancer. A new peer mental-wellness support program, called Color Cancer Connect (CCC) supports cancer patients, survivors and their caregivers by teaching them evidence-based skills to manage the emotional impact of cancer. This study will examine all three programs (i.e., patient, survivor, caregiver) to gather data to measure the impact of the program on emotional well-being, quality of life and health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Lived experience as either a current cancer patient, cancer survivor or caregiver of someone with cancer
* Adult - 18+
* Has health insurance provided by employer or union (can be dependent of person on insurance)
* Read/speak English
* Have access to internet and personal email account

Exclusion Criteria:

* Severe mental illness that is disruptive to other group members

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-01-25 (Actual)

PRIMARY OUTCOMES:
Depression | Multiple time points across 8 months (waitlist; baseline, 2 months post waitlist, 3 months post waitlist, 2 months post program start, 3 months post program start) or 5 months (intervention; baseline, 2 months post program start, 3 months post program)
  Patient Health Questionnaire-9 (PHQ-9)

CONTACTS AND LOCATIONS:
Locations (1):
- Color Health, Burlingame, California, United States

IPD SHARING:
Plan to Share IPD: Undecided